CLINICAL TRIAL: NCT01254929
Title: 18F-Fluoride PET Bone Scans Versus Traditional 99mTc-MDP Gamma Camera Bone Scans for the Diagnosis of Bone Metastases: a Blinded, Prospective Trial
Brief Title: F-18 PET Bone Scans Versus Tc-99m Bone Scans for the Diagnosis of Bone Metastases
Status: Completed | Type: Observational
Sponsor: Seattle Nuclear Medicine (Other)
Responsible Party: Principal Investigator, David Djang, Nuclear medicine physician, Seattle Nuclear Medicine
Other Study IDs: CAG00065R
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Cancer; Bone Metastases
Keywords: Cancer; Bone metastases
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- F-18 PET bone scan group: Patients with a diagnosis of cancer and clinical concern for bone metastases. They will undergo an F-18 PET bone scan for diagnostic imaging.
  Interventions: Device: F-18 PET bone scan
- Tc-99m MDP bone scan group: Patients with a diagnosis of cancer and clinical concern for bone metastases. They will undergo a Tc-99m MDP bone scan for diagnostic imaging.
  Interventions: Device: Tc-99m bone scan

INTERVENTIONS:
Device: F-18 PET bone scan — Following the intravenous administration of approximately 10 mCi F-18, subjects will undergo an F-18 PET bone scan.
  Other Names: PET Allegro scanner
  Groups: F-18 PET bone scan group
Device: Tc-99m bone scan — Following the intravenous administration of approximately 30mCi Tc-99m MDP, subjects will undergo a traditional bone scan on a gamma camera.
  Other Names: Philips/ADAC Genesys gamma camera
  Groups: Tc-99m MDP bone scan group

SUMMARY:
The purpose of this study is to compare 18F-Fluoride PET bone scans to traditional 99mTc-MDP bone scan to determine if one is better for diagnosing bone metastases.

DETAILED DESCRIPTION:
Compare the diagnostic sensitivity, specificity, and accuracy of 18F-Fluoride PET bone scans versus traditional 99mTc-MDP bone scans for detecting bone metastases.

Determine if there is a significant change in clinical management between the two types of scans.

Measure and compare the number of equivocal or uncertain findings that would have caused additional testing, particularly additional imaging studies, to be performed for confirmation when using 18F-Fluoride PET bone scans versus 99mTc-MDP bone scans.

To quantify any adverse events resulting from either scan.

To perform subgroup analyses according to cancer cell type.

ELIGIBILITY:
Inclusion Criteria:

* Patient has cancer
* Has been referred for evaluation of bone metastases
* Patient or patient's legal representative can understand and consent to enrollment in the study
* Must be 18 years or older
* Can remain still during the scan (approximately one hour)
* Patient has Medicare

Exclusion Criteria:

* Patient does not have Medicare
* Under the age of 18
* Cannot lie still for the necessary time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have cancer and have been referred for evaluation for bone metastases.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Accurate identification of bone metastases | Upon study completion (2-3 years)
  Individual subjects will be reviewed 6-12 months after their bone scans, utilizing all clinical and imaging data available, to determine diagnostic accuracy of each bone scan.

SECONDARY OUTCOMES:
Change in clinical management | Upon study completion (2-3 years)
  We will be sending out clinical questionnaires to the referring physicians, asking if the bone scan results helped and/or changed their clinical management. Cumulative data for each type of bone scan will be compared.
Determine if F-18 PET bone scans lead to fewer follow-up imaging studies. | Upon study completion (2-3 years)
  The Tc-99m bone scans often give equivocal results that require other imaging studies, such as CT or MRI, for further evaluation. F-18 PET bone scans may give more definitive interpretations, and thus may lead to fewer follow-up studies being recommended/obtained.
Quantify any adverse events from either type of scan. | Upon study completion (2-3 years)
  Any adverse events related to either type of scan will be recorded. Adverse events would be rare.
Perform subgroup analyses according to cancer cell type. | Upon study completion (2-3 years)
  Both types of bone scans may be more or less accurate depending on the cancer cell type. We will attempt to address that question by performing subgroup analyses.

CONTACTS AND LOCATIONS:
Overall Officials: David Djang, MD, Principal Investigator — Seattle Nuclear Medicine
Locations (1):
- Seattle Nuclear Medicine, Seattle, Washington, United States